CLINICAL TRIAL: NCT07361302
Title: TENACITY - A Phase III, Prospective, Randomized, Open-label, Blinded Endpoint Assessment (PROBE) to Assess Efficacy and Safety of i.v. Tenecteplase vs Standard of Care in Patients With Acute Ischemic Stroke (Including Wake-up Stroke), Last Known Well >4.5 h With Imaging Evidence of Salvageable Ischemic Tissue
Brief Title: A Study to Test if Tenecteplase Helps People to Recover From an Acute Stroke When Given More Than 4.5 Hours After the Person Was Last Seen Well
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1123-0060; 2025-522542-40-00 (EU CTIS Number); U1111-1323-6001 (Registry Identifier: WHO - International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2026-01-14; First posted 2026-01-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenecteplase treatment arm (Experimental)
  Interventions: Drug: Tenecteplase
- Standard of care treatment arm (Active Comparator)
  Interventions: Drug: Standard of care treatment

INTERVENTIONS:
Drug: Tenecteplase — Tenecteplase
  Arms: Tenecteplase treatment arm
Drug: Standard of care treatment — Standard of care treatment
  Arms: Standard of care treatment arm

SUMMARY:
This study is open to adults who had an acute stroke caused by a clot blocking a blood vessel in the brain (acute ischemic stroke). This study is for people who had an acute stroke or woke up with a stroke and were last seen well more than 4.5 hours before joining the study. Participants need to have imaging that shows there is brain tissue that can still be saved. They also should not be planned to receive a procedure to remove the blood clot.

The purpose of this study is to find out whether a medicine called tenecteplase helps people recover from an acute stroke. Tenecteplase is already used to treat people within 4.5 hours after they had a stroke. This study tests if tenecteplase also helps if it is given more than 4.5 hours after the stroke.

Participants are put into 2 groups randomly, which means by chance. One group gets tenecteplase as a single injection into a vein. The other group receives standard medical practice. Participants have an equal chance of receiving tenecteplase or the standard treatment.

Participants are in the study for about 3 months. In the beginning, participants stay in the hospital for about 1 week. During the study, participants have 7 clinical examinations or visits. The last 2 of these visits will likely be done from home, allowing participants to complete certain assessments remotely. Doctors regularly test participants' recovery using a scale that measures the level of disability or dependence in daily activities. The results are compared between the 2 groups to see whether the treatment works. The doctors also check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria:

1. Male or female ≥18 years old and at least at the legal age of consent in countries where it is greater than 18 years
2. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
3. Acute ischaemic stroke (including wake-up stroke) affecting the supratentorial circulation (anterior cerebral artery (ACA), middle cerebral artery (MCA), and posterior cerebral arteries (PCA)) last known well >4.5 h before time of presumed randomisation
4. Pre-stroke modified Rankin scale (mRS) ≤1
5. Imaging eligibility by magnetic resonance imaging (MRI)computed tomography (CT)

Exclusion criteria:

1. Intention to proceed to mechanical thrombectomy (MT) at the same site (hospital) of randomisation
2. Occlusion of the internal carotid artery (ICA)
3. High-risk patients (increased risk of thrombolysis related hemorrhage)
4. Any intracranial hemorrhage detected on non-contrast computed tomography (NCCT) or MRI scans
5. Contra-indication to contrast brain imaging with CT and MRI
6. Severe stroke as assessed clinically (National Institute of Health Stroke Scale (NIHSS) > 25)
7. Non-disabling minor stroke symptoms (NIHSS ≤5), or rapidly improving symptoms at the discretion of the investigator
8. Imaging or clinical findings not indicative of acute ischemic stroke or suggesting stroke older than 72 h
9. Patients scheduled to receive intravenous (i.v.) thrombolysis as standard of care Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1325 (Estimated)
Dates: Start 2026-02-17 (Estimated); Primary Completion 2027-10-02 (Estimated); Study Completion 2027-10-02 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) score of 0-1 at Day 90 | at day 90
  The Modified Rankin Scale, MRS, is a tool used to evaluate disability after a stroke. The score ranges from 0 to 6, with higher values indicating greater severity of the disability.

SECONDARY OUTCOMES:
mRS (ordinal) at Day 90 | at day 90
Early neurological improvement (reduction in acute - 24-hour National Institute of Health Stroke Scale (NIHSS) score of ≥8 or value of 0/1) | at baseline/randomisation, 24 hours after randomization
  NIHSS is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. It is composed of 11 items. The score ranges from 0 to a maximum of 42. For each item a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment.
mRS 0-2 at Day 90 | at Day 90
Symptomatic intracranial haemorrhage (sICH) as defined by Safety Implementation of Thrombolysis in Stroke: Monitoring Study (SITS-MOST) criteria at 36 h | after 36 hours
sICH as defined by European Cooperative Acute Stroke Study (ECASS) III criteria at 36 h | after 36 hours
Death from any cause within 90 days | up to 90 days

CONTACTS AND LOCATIONS:
Locations (181):
- Argentina (15):
  - Sanatorio Güemes, Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma Buenos Aires
  - CEMIC, Ciudad Autonoma Buenos Aires
  - Hospital General de Agudos Dr. J. M. Ramos Mejia, Ciudad Autonoma Buenos Aires
  - Fundacion para la Lucha contra las Enfermedades Neurologicas de la Infancia - FLENI, Ciudad Autonoma Buenos Aires
  - Complejo Medico de la Policia Federal Argentina Churruca Visca, Ciudad Autonoma Buenos Aires
  - Clinica Privada Velez Sarfield, Córdoba
  - Nuevo Hospital San Roque, Córdoba
  - Sanatorio Allende, Córdoba
  - Sanatorio Privado Duarte Quiros De Clinica Colombo SA, Córdoba
  - Sanatorio de la Canada, Córdoba
  - Hospital Cordoba, Córdoba
  - Hospital Privado de Comunidad, Mar del Plata
  - Hospital Universitario Austral, Pilar
  - Hospital Privado de Rosario, Rosario
- Australia (7):
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Eastern Health-Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Bulgaria (15):
  - MHAT "Puls" AD, Blagoevgrad
  - MHAT Heart and brain, Burgas
  - MHAT Sv. Ivan Rilski EOOD, Gorna Oryahovitsa
  - MHAT City Clinic Saint Georgi Ltd, Montana
  - MHAT Heart and brain, Pleven
  - University Multiprofile Hospital For Active Treatment Dr. Georgi Stranski EAD, Pleven
  - UMHAT "Kaspela", EOOD, Plovdiv
  - UMHAT "Sv. Georgi", EAD, Plovdiv
  - UMHAT "Medika Ruse" OOD, Rousse
  - MHAT "Hadzhi Dimitar" OOD, Silven
  - MHATNP "Sv. Naum" EAD, Sofia
  - University First MHAT-Sofia "St. Joan Krastitel" EAD, Sofia
  - Acibadem City Clinic Tokuda University Hospital EAD, Sofia
  - Multiprofile Hospital MHATEM 'Pirogov', Sofia, Sofia
  - University Hospital St. Anna, Sofia
- China (33):
  - The People's Hospital of Anyang City, Anyang
  - Baoji Central Hospital, Baoji
  - Inner Mongolia Baogang Hospital, Baotou
  - Cap Med University, Beijing
  - Peking University Third Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Hunan Province People's Hospital (The First Affiliated Hospital of Hunan Normal University), Changsha
  - Chifeng Traditional Chinese and Mongolian Medicine Hospital, Chifeng
  - Daqing Oilfield General Hospital, Daqing
  - General Hospital of Fushun Mining Bureau, Fushun
  - Third Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The Second Hospital of Harbin Medical University, Haerbin
  - The First Affiliated Hospital of University of South China, Hengyang
  - Meihekou Central Hospital, Jilin
  - Jinhua Municipal Central Hospital, Jinhua
  - First People's hospital of Yunann Province, Kunming
  - Liaocheng People's Hospital, Liaocheng
  - Linfen Central Hospital, Linfen
  - Linyi People's Hospital, Linyi
  - The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - Nanyang Central Hospital, Nanyang
  - Pingxiang People's Hospital, Pingxiang
  - Qingdao Municipal Hospital, Qingdao
  - Huashan Hospital, Fudan University, Shanghai
  - Affiliated Central Hospital of Shenyang Medical College, Shenyang
  - Shanxi Cardiovascular Hospital, Taiyuan
  - The First People's Hospital of Tancheng, Tengzhou
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - The Central Hospital of Wuhan, Wuhan
  - The People's Hospital Of Xuancheng City, Xuancheng
  - Xuzhou Central Hospital, Xuzhou
  - Zigong No. 1 People's Hospital, Zigong
- Greece (11):
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - Athens Euroclinic S.A., Athens
  - Athens Naval Hospital, Athens
  - Eginitio Hospital, Athens
  - University General Hospital Attikon, Athens
  - Metropolitan Hospital, Athens, Neo Faliro
  - University General Hospital of Heraklion, Heraklion
  - General University Hospital of Larissa, Larissa
  - General University Hospital of Patras, Pátrai
  - University General Hospital of Thessaloniki AHEPA, Thessaloniki
  - General Hospital Of Thessaloniki Papageorgiou, Thessaloniki
- Hungary (8):
  - Semmelweis University, Budapest
  - Budapesti Uzsoki Utcai Korhaz, Budapest
  - Pest Megyei Flor Ferenc Hospital, Kistarcsa
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz, Nyíregyháza
  - University of Pecs, Pécs
  - University of Szeged, Szeged
  - Fejer Varmegyei Szent Gyoergy Egyetemi Oktato Korhaz, Székesfehérvár
- India (23):
  - Zydus Hospital - Ahmedabad, Ahmedabad
  - Bangalore Medical College, Bangalore
  - KLES Dr. Prabhakar Kore Hospital and Medical Research Centre, Belagavi
  - S.P. Medical College & Associated Group of Hospitals, Bikaner
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - K.G. Hospital and Post Graduate Medical Institute, Coimbatore
  - Lalitha Super Speciality Hospital, Guntur
  - Yashoda Hospitals, Somajiguda, Hyderabad
  - Institute of Neurosciences Kolkata, Kolkata
  - Bangur Institute of Neurosciences, Kolkata
  - Christian Medical College, Ludhiana, Ludhiana
  - Chopda Medicare and Research Centre Pvt Ltd, Nashik
  - BLK-Max Super Speciality Hospital, Delhi, New Delhi
  - Max Super Speciality Hospital, New Delhi
  - Deenanath Mangeshkar Hospital and Research Centre, Pune
  - Synergy Superspeciality Hospital, Rajkot
  - Bhaktivedanta Hospital & Research Institute, Thane
  - Sree Chitra Tirunal Institute for Medical Sciences & Technology, Thiruvananthapuram
  - City Neurology Centre, Varanasi
  - Christian Medical College, Vellore, Vellore
  - Government Siddhartha Medical College, Vijayawada
  - Visakha Institute of Medical Sciences, Visakhapatnam
  - Government Medical College Vizianagaram, Vizianagaram
- Indonesia (10):
  - Siloam Hospitals Denpasar, Badung
  - Immanuel Hospital Bandung, Bandung
  - Dr. Cipto Mangunkusumo Hospital, Jakarta
  - Siloam Hospitals TB Simatupang, Jakarta
  - Mahar Mardjono National Brain Center Hospital, Jakarta
  - Airlangga University Hospital, Surabaya
  - Siloam Hospitals Lippo Village, Tangerang
  - Bethesda Hospital, Yogyakarta
  - RS Akademik UGM, Yogyakarta
  - Sardjito Hospital, Yogyakarta
- Kazakhstan (2):
  - City Multidisciplinary Hospital No 2, Astana
  - National Coordination Center for Emergency Medicine, Astana
- Malaysia (4):
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Universiti Sains Malaysia, Kota Bharu
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Universiti Putra Malaysia, Serdang
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Sykehuset Ostfold HF, Grålum
  - Helse Stavanger, Stavanger Universitetssykehus, Stavanger
- Romania (6):
  - Spitalul Clinic Județean De Urgența Arad, Arad
  - Spitalul Clinic Judetean de Urgenta Brasov, Brasov
  - Spitalul Clinic Judetean De Urgenta Sfantul Apostol Andrei Constanta, Constanța
  - Spitalul Judetean de Urgenta Piatra Neamt, Piatra Neamţ
  - Spitalul Judetean De Urgenta Sfantul Ioan Cel Nou Suceava, Suceava
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Mureş
- Spain (17):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron - VHIR, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Ruber Juan Bravo, Madrid
  - Hospital Universitario De La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen De La Macarena, Seville
  - Hospital Universitari Mutua de Terrasa, Terrassa
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (8):
  - Chang Gung Memorial Hospital Chiayi, Buzi
  - Chang Gung Memorial Hospital-Keelung, Keelung
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- Thailand (8):
  - Phramongkutklao Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Thammasat University Hospital, Klong Luang
  - Lampang Hospital, Lampang
  - Sunprasitthiprasong Hospital, Muang
- Vietnam (11):
  - Da Nang Hospital, Da Nang
  - Viet Tiep Hospital, Haiphong
  - Bach Mai hospital, Hanoi
  - Le Van Thinh Hospital, Ho Chi Minh City
  - Military Hospital 175, Ho Chi Minh City
  - Nguyen Tri Phuong Hospital, Ho Chi Minh City
  - Nhan Dan Gia Dinh Hospital, Ho Chi Minh City
  - People's Hospital 115, Ho Chi Minh City
  - Thong Nhat Hospital HCMC, Ho Chi Minh City
  - University Medical Center HCMC, Ho Chi Minh City
  - Phu Tho General Hospital, Việt Trì

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a "Document Sharing Agreement". For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com